CLINICAL TRIAL: NCT02898636
Title: Identification of Protein Markers of Vitality in Skin Wounds by Forensic Multiplex Analysis
Brief Title: Identification of Biomarkers in the Legal Medical Skin Wounds
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9552
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Legal Medical Skin Wounds
MeSH Terms: interventions — Autopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: autopsy — At autopsy achieving adequate sampling of lesions and healthy skin

SUMMARY:
Identify the cytokine or combination of cytokines, with the best diagnostic performance to characterize the vital nature of a skin wound in the body.

DETAILED DESCRIPTION:
Determining the vitality of skin wounds, that is to say their antemortem character, is an important issue in forensic pathology. The only criterion vitality currently recognized (but whose diagnostic performance remains limited) is the microscopic demonstration of an inflammatory infiltrate of neutrophils. The search for more reliable diagnostic biomarkers is required. By their early expression of the injury site, inflammatory cytokines are potential candidates and their quantification in injured skin could optimize the diagnosis of vitality injury.

The objective is to identify the cytokine or combination of cytokines, with the best diagnostic performance to characterize the vital nature of a skin wound in the body.

ELIGIBILITY:
Inclusion Criteria:

* Adult died 18 years or more
* Having at least one recent ante-mortem skin wound (occurring less than 4 hours prior to death)
* Hours of death and the establishment of the ante-mortem wound known (date, hours and minutes)

Exclusion Criteria:

* Immunocompromised patients (HIV infection, immunosuppressive therapy ...)
* Putrefaction signs (abdominal patch of green ...)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient undergoing a forensic autopsy
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
measures cytokines | 1 day
  multiplex analysis electrochemoluminescence: Six cytokines candidates selected from a literature review (IFN-γ, IL-1β, IL-6, IL-10, IL-12 p70, TNF-α) will be assayed in conjunction with the MSD technology (V-PLEX proinflammatory Panel 1 human Kit) after tissue extraction and determination of total protein concentration in each sample.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Antoine PEYRON, MD, Study Director — University Hospital, Montpellier
Locations (1):
- PEYRON, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided